CLINICAL TRIAL: NCT04761861
Title: Vildagliptin for Treatment of Antipsychotic-induced Dyslipidemia: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Vildagliptin for Treatment of Antipsychotic-induced Dyslipidemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2021NEUR
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Dyslipidemias
MeSH Terms: conditions — Schizophrenia; Dyslipidemias | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vildagliptin (Experimental): Vildagliptin 50 mg tablet daily
  Interventions: Drug: Vildagliptin 50 MG
- Placebo (Placebo Comparator): Placebo tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin 50 MG — Vildagliptin 50 MG tablet once daily
  Arms: Vildagliptin
Drug: Placebo — Placebo one tablet daily
  Arms: Placebo

SUMMARY:
Almost all antipsychotics can induce dyslipidemia, but no treatment has been established. Vildagliptin can improve lipid levels in obese patients. The investigators conducted a randomized, placebo-controlled study to test the efficacy of vildagliptin for antipsychotic-induced dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorder-Fourth Edition (DSM-Ⅳ) criteria for schizophrenia dyslipidemia after antipsycotic treatment the duration of illness was less than 12 months taking only one antipsychotic stable outpatient the total score of Positive and Negative Syndrome Scale (PANSS)≤60.

Exclusion Criteria:

* liver or renal diseases pregnant or lactating women cardiovascular diseases hypertension or diabetes mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
low-density lipoprotein cholesterol | week 12
  low-density lipoprotein cholesterol

SECONDARY OUTCOMES:
high-density lipoprotein cholesterol | week 12
  high-density lipoprotein cholesterol
Serum stem cell growth factor beta | week 12
  Serum stem cell growth factor beta
FAM19A5 serum level | 12 weeks
  FAM19A5 serum level
TNF-alpha serum level | 12 weeks
  TNF-alpha serum level
Adverse drug reactions | 12 weeks
  Adverse drug reactions

OTHER OUTCOMES:
body mass index | 12 weeks
  body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF